CLINICAL TRIAL: NCT01104662
Title: A Prospective, Multicenter, Randomized, Evaluator-blinded, Comparator-controlled Study to Describe the Safety and Efficacy of Daptomycin for the Treatment of Complicated Skin and Skin Structure Infections (cSSSI) and Staphylococcus Aureus Bacteremia Among Subjects With Moderate or Severe Renal Impairment
Brief Title: Study of Daptomycin Safety and Efficacy for Complicated Skin and Skin Structure Infections (cSSSI) and Bacteremia in Renal Impairment
Acronym: RENSE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Cubist has reached an agreement with the FDA that enrollment in the DAP-RENSE-08-05 study can stop.
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3009-022; DAP-RENSE-08-05 (Other: Cubist Study Number)
Record Dates: First submitted 2010-04-02; First posted 2010-04-15 (Estimated); Results first posted 2015-05-13 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Complicated Skin and Skin Structure Infections; S. Aureus Bacteremia; Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — Vancomycin; Daptomycin; Nafcillin; Oxacillin; Cloxacillin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Daptomycin, Bacteremia, Severe Renal Impairment (Experimental): Cohort 1. Daptomycin was given intravenously 6 milligrams per kilogram (mg/kg) per administration. For bacteremia participants with Creatinine Clearance (CLcr) below 30 milliliters per minute (mL/min) and currently receiving hemodialysis, daptomycin was administered immediately following each hemodialysis session (3 per week) for 14 to 42 days based on disease resolution or Investigator discretion. For participants not receiving dialysis, daptomycin was administered every 48 hours for 14 to 42 days based on disease resolution or Investigator discretion.
  Interventions: Drug: Daptomycin
- Vancomycin or SSP, Bacteremia, Severe Renal Impairment (Active Comparator): Cohort 1. Participants randomized to the comparator therapy group received vancomycin or penicillinase-resistant penicillin (nafcillin, oxacillin, or cloxacillin). Investigators were allowed to select an agent based on local availability and normal treatment practices. Participants randomized to comparator subsequently found to have an infection caused by Methicillin-Susceptible Staphylococcus Aureus (MSSA) could have switched from vancomycin to penicillinase-resistant penicillin (nafcillin, oxacillin, or cloxacillin) at the Investigator's discretion. All treatments were dosed per Investigator's discretion and were administered intravenously (IV) until end of antibiotic therapy for bacteremia or until hospital discharge, whichever occurred first. Investigators treated participants according to their usual decision-making and discretion.
  Interventions: Drug: Vancomycin; Drug: Semi-Synthetic Penicillin
- Daptomycin, Bacteremia, Moderate Renal Impairment (Experimental): Cohort 2. Daptomycin was given intravenously 6 milligrams per kilogram (mg/kg) per administration. For bacteremia participants with CLcr values between 30 and 50 mL/min not receiving dialysis, daptomycin was administered every 24 hours for 14 to 42 days based on disease resolution or Investigator discretion.
  Interventions: Drug: Daptomycin
- Vancomycin or SSP , Bacteremia, Moderate Renal Impairment (Active Comparator): Cohort 2. Participants randomized to the comparator therapy group received vancomycin or penicillinase-resistant penicillin (nafcillin, oxacillin, or cloxacillin). Investigators were allowed to select an agent based on local availability and normal treatment practices. Participants randomized to comparator subsequently found to have an infection caused by MSSA could have switched from vancomycin to penicillinase-resistant penicillin (nafcillin, oxacillin, or cloxacillin) at the Investigator's discretion. All treatments were dosed per Investigator's discretion and were administered IV until end of antibiotic therapy for bacteremia or until hospital discharge, whichever occurred first. Investigators treated participants according to their usual decision-making and discretion.
  Interventions: Drug: Vancomycin; Drug: Semi-Synthetic Penicillin
- Daptomycin, cSSSI, Severe Renal Impairment (Experimental): Cohort 3. Daptomycin was given intravenously 4 milligrams per kilogram (mg/kg) per administration. For cSSSI participants with CLcr below 30 mL/min and currently receiving hemodialysis, daptomycin was administered immediately following each hemodialysis session (3 per week) for 7 to 14 days based on disease resolution or Investigator discretion. For participants not receiving dialysis, daptomycin was administered every 48 hours for 7 to 14 days based on disease resolution or Investigator discretion.
  Interventions: Drug: Daptomycin
- Vancomycin or SSP , cSSSI, Severe Renal Impairment (Active Comparator): Cohort 3. Participants randomized to the comparator therapy group received vancomycin or penicillinase-resistant penicillin (nafcillin, oxacillin, or cloxacillin). Investigators were allowed to select an agent based on local availability and normal treatment practices. Participants randomized to comparator subsequently found to have an infection caused by MSSA could have switched from vancomycin to penicillinase-resistant penicillin (nafcillin, oxacillin, or cloxacillin) at the Investigator's discretion. All treatments were dosed per Investigator's discretion and were administered IV until end of antibiotic therapy for cSSSI or until hospital discharge, whichever occurred first. Investigators treated participants according to their usual decision-making and discretion.
  Interventions: Drug: Vancomycin; Drug: Semi-Synthetic Penicillin
- Daptomycin, cSSSI, Moderate Renal Impairment (Experimental): Cohort 4. Daptomycin was given intravenously 4 milligrams per kilogram (mg/kg) per administration. For cSSSI participants with CLcr values between 30 and 50 mL/min not receiving dialysis, daptomycin was administered every 24 hours for 7 to 14 days based on disease resolution or Investigator discretion.
  Interventions: Drug: Daptomycin
- Vancomycin or SSP , cSSSI, Moderate Renal Impairment (Active Comparator): Cohort 4. Participants randomized to the comparator therapy group received vancomycin or penicillinase-resistant penicillin (nafcillin, oxacillin, or cloxacillin). Investigators were allowed to select an agent based on local availability and normal treatment practices. Participants randomized to comparator subsequently found to have an infection caused by MSSA could have switched from vancomycin to penicillinase-resistant penicillin (nafcillin, oxacillin, or cloxacillin) at the Investigator's discretion. All treatments were dosed per Investigator's discretion and were administered IV until end of antibiotic therapy for cSSSI or until hospital discharge, whichever occurred first. Investigators treated participants according to their usual decision-making and discretion.
  Interventions: Drug: Vancomycin; Drug: Semi-Synthetic Penicillin

INTERVENTIONS:
Drug: Vancomycin
  Arms: Vancomycin or SSP , Bacteremia, Moderate Renal Impairment; Vancomycin or SSP , cSSSI, Moderate Renal Impairment; Vancomycin or SSP , cSSSI, Severe Renal Impairment; Vancomycin or SSP, Bacteremia, Severe Renal Impairment
Drug: Daptomycin
  Other Names: Cubicin
  Arms: Daptomycin, Bacteremia, Moderate Renal Impairment; Daptomycin, Bacteremia, Severe Renal Impairment; Daptomycin, cSSSI, Moderate Renal Impairment; Daptomycin, cSSSI, Severe Renal Impairment
Drug: Semi-Synthetic Penicillin
  Other Names: SSP, nafcillin, oxacillin, cloxacillin
  Arms: Vancomycin or SSP , Bacteremia, Moderate Renal Impairment; Vancomycin or SSP , cSSSI, Moderate Renal Impairment; Vancomycin or SSP , cSSSI, Severe Renal Impairment; Vancomycin or SSP, Bacteremia, Severe Renal Impairment

SUMMARY:
This is a multicenter, randomized, evaluator-blinded, comparator-controlled study. Participants were to be randomized (1:1) to daptomycin or comparator, stratified by degree of renal impairment (creatinine clearance [CLcr] 30 - 50 milliliters per minute [mL/min] [moderate impairment] and <30 mL/min [severe impairment]) and by type of infection (bacteremia and complicated skin and skin structure infections [cSSSI]) to create 4 cohorts defined as follows:

* Cohort 1: Bacteremia and CLcr <30 mL/min
* Cohort 2: Bacteremia and CLcr 30 - 50 mL/min
* Cohort 3: cSSSI and CLcr <30 mL/min
* Cohort 4: cSSSI and CLcr 30 - 50 mL/min

Participants will be treated and evaluated for safety and microbiological and clinical efficacy in accordance with their type of infection and degree of renal impairment. Peak and trough samples will be collected to assess exposure to daptomycin for participants on Day 1 and following the 5th dose.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or female ≥18 years of age
* Diagnosis of cSSSI or Staphylococcus aureus (S. aureus) bacteremia
* Renal impairment of CLcr of 30 - 50 mL/min or CLcr <30 mL/min per Cockcroft-Gault equation using actual body weight
* Functioning hemodialysis access and on stable regimen for those receiving dialysis
* In appropriate health for the study with no acute or chronic illnesses that could adversely impact safety or ability to complete the study

Specific inclusion criteria for cSSSI:

* Presence of a wound infection, major abscess, severe carbunculosis, infected ulcers, dialysis access site infection, or other type of infection in presence of complicating factor
* At least 3 of the following symptoms, signs, or laboratory values of a skin infection: elevated temperature; elevated white blood cell (WBC) count; pain; tenderness; swelling; erythema greater than 1 centimeter (cm) beyond wound edge; induration; pus formation
* Evidence of a Gram-positive infecting pathogen as indicated by positive Gram stain or culture obtained within 96 hours prior to study drug administration
* Infection of sufficient severity to require parenteral antimicrobial therapy

Specific inclusion criteria for S. aureus bacteremia:

• Documented S. aureus bacteremia defined as at least one positive blood culture for S. aureus obtained within 96 hours prior to the first dose of study medication

Exclusion Criteria:

* Pregnant or lactating females, or unwilling to practice barrier methods of birth control
* Received an investigational drug (including experimental biologic agents) within 30 days of study entry
* Unable to discontinue use of HMG-CoA reductase inhibitor therapy while on study
* Known allergy or intolerance to daptomycin, penicillin, or vancomycin
* Active intravenous (IV) drug abuse
* Confirmed or suspected osteomyelitis, septic arthritis, meningitis, epidural abscess, intra-abdominal infection, pneumonia, or infective endocarditis
* Required use of non-study systemic antibacterial agent with activity against target pathogen
* History of muscular disease
* Neurological disease except stroke >6 months prior to study entry
* Intramuscular injection within 7 days of study drug administration
* Moribund clinical condition (high likelihood of death during next 3 days)
* Shock or hypotension (supine systolic blood pressure <80 millimeters of mercury [mmHg])
* Body mass index (BMI) <18 or >40 kilograms per meter squared (kg/m^2) [BMI = weight (kg)/height (m^2)]
* Known human immunodeficiency virus (HIV) infection with CD4 count ≤200 cells/millimeter (mm)^3
* Neutropenic participants with an absolute neutrophil count ≤500 cells/mm^3
* Anticipated to develop neutropenia absolute neutrophil count ≤500 due to prior or planned chemotherapy
* Alanine aminotransferase (ALT) value >3 × upper limit of normal (ULN)
* Aspartate aminotransferase (AST) value >3 × ULN
* Total bilirubin values ≥ 1.5 x ULN associated with ALT values >3 x ULN
* Creatine phosphokinase (CPK) value >2 × ULN
* Hemoglobin <8 grams per deciliter (gm/dL)
* Unlikely to comply with study procedures or to return for evaluations
* History of rhabdomyolysis
* Prior enrollment into this study
* Infections caused by Gram-positive pathogens known to be resistant to daptomycin or selected comparator agent

Specific exclusion criteria for cSSSI:

* Minor or superficial skin infections as the primary site of infection
* Cellulitis or erysipelas not associated with complicating factor as primary site of infection
* Perirectal abscess, hidradenitis suppurativa, concomitant gangrene, myositis, multiple infected ulcers at distant sites, necrotizing fasciitis, or infected third-degree burn wounds
* Infections requiring emergency surgery
* Infections suspected or documented to be due exclusively to gram-negative, anaerobic, or fungal organism
* Confirmed or suspected disorder that could interfere with the evaluations (for example, primary skin disorders)
* Use of a topical antibiotic at the site of the infection
* Use of systemic antibacterial therapy for the infection for >24 hours within 48 hours prior to start of study drug unless (a) infecting Gram-positive pathogen resistant to therapy or (b) therapy administered for 3 or more days with worsening or no improvement
* Planned surgical treatment that is considered curative of the infection

Specific exclusion criteria for S. aureus bacteremia:

* Has intravascular foreign material at the time the positive blood culture was drawn (for example., intracardiac pacemaker wires, percutaneous or implanted venous catheters, vascular grafts) unless material removed within 4 days after first dose of study medication or approval of medical monitor (exceptions: vascular stents in place for >6 months, permanent pacemaker attached via epicardial leads, or any dialysis access device unless this material is felt to be infected)
* Prosthetic heart valve
* Cardiac decompensation or valve damage or both with high likelihood of valve surgery in the 3 days after randomization
* Polymicrobial blood infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-04-19 (Actual); Primary Completion 2012-06-12 (Actual); Study Completion 2012-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellie Hershberger, Pharm.D., Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (10):
- United States (10):
  - Azusa, California
  - Los Angeles, California
  - Torrance, California
  - Washington D.C., District of Columbia
  - Decatur, Georgia
  - Somers Point, New Jersey
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - West Reading, Pennsylvania
  - Mission, Texas

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Vancomycin or SSP, Bacteremia, Severe Renal Impairment: Cohort 1. Participants randomized to the comparator therapy group received vancomycin or penicillinase-resistant penicillin/semi-synthetic penicillin (SSP; for example, nafcillin, oxacillin, or cloxacillin). Investigators were allowed to select an agent based on local availability and normal treatment practices. Participants randomized to comparator subsequently found to have an infection caused by Methicillin-Susceptible Staphylococcus Aureus (MSSA) could have switched from vancomycin to penicillinase-resistant penicillin (nafcillin, oxacillin, or cloxacillin) at the Investigator's discretion. All treatments were dosed per investigator's discretion and were administered intravenously until end of antibiotic therapy for bacteremia or until hospital discharge, whichever occurred first. Investigators treated participants according to their usual decision-making and discretion.
- Vancomycin or SSP, Bacteremia, Moderate Renal Impairment: Cohort 2. Participants randomized to the comparator therapy group received vancomycin or penicillinase-resistant penicillin (nafcillin, oxacillin, or cloxacillin). Investigators were allowed to select an agent based on local availability and normal treatment practices. Participants randomized to comparator subsequently found to have an infection caused by MSSA could have switched from vancomycin to penicillinase-resistant penicillin (nafcillin, oxacillin, or cloxacillin) at the Investigator's discretion. All treatments were dosed per investigator's discretion and were administered IV until end of antibiotic therapy for bacteremia or until hospital discharge, whichever occurred first. Investigators treated participants according to their usual decision-making and discretion.
- Daptomycin, cSSSI, Severe Renal Impairment: Cohort 3. Daptomycin was given intravenously 4 milligrams per kilogram (mg/kg) per administration. For complicated skin and skin structure infections (cSSSI) participants with CLcr below 30 mL/min and currently receiving hemodialysis, daptomycin was administered immediately following each hemodialysis session (3 per week) for 7 to 14 days based on disease resolution or Investigator discretion. For participants not receiving dialysis, daptomycin was administered every 48 hours for 7 to 14 days based on disease resolution or Investigator discretion.
- Vancomycin or SSP, cSSSI, Severe Renal Impairment: Cohort 3. Participants randomized to the comparator therapy group received vancomycin or penicillinase-resistant penicillin (nafcillin, oxacillin, or cloxacillin). Investigators were allowed to select an agent based on local availability and normal treatment practices. Participants randomized to comparator subsequently found to have an infection caused by MSSA could have switched from vancomycin to penicillinase-resistant penicillin (nafcillin, oxacillin, or cloxacillin) at the Investigator's discretion. All treatments were dosed per investigator's discretion and were administered IV until end of antibiotic therapy for cSSSI or until hospital discharge, whichever occurred first. Investigators treated participants according to their usual decision-making and discretion.
- Vancomycin or SSP, cSSSI, Moderate Renal Impairment: Cohort 4. Participants randomized to the comparator therapy group received vancomycin or penicillinase-resistant penicillin (nafcillin, oxacillin, or cloxacillin). Investigators were allowed to select an agent based on local availability and normal treatment practices. Participants randomized to comparator subsequently found to have an infection caused by MSSA could have switched from vancomycin to penicillinase-resistant penicillin (nafcillin, oxacillin, or cloxacillin) at the Investigator's discretion. All treatments were dosed per investigator's discretion and were administered IV until end of antibiotic therapy for cSSSI or until hospital discharge, whichever occurred first. Investigators treated participants according to their usual decision-making and discretion.
Period: Overall Study
Arm/Group | Daptomycin, Bacteremia, Severe Renal Impairment | Vancomycin or SSP, Bacteremia, Severe Renal Impairment | Daptomycin, Bacteremia, Moderate Renal Impairment | Vancomycin or SSP, Bacteremia, Moderate Renal Impairment | Daptomycin, cSSSI, Severe Renal Impairment | Vancomycin or SSP, cSSSI, Severe Renal Impairment | Daptomycin, cSSSI, Moderate Renal Impairment | Vancomycin or SSP, cSSSI, Moderate Renal Impairment
Started | 20 | 21 | 5 | 4 | 15 | 16 | 5 | 6
Received at Least 1 Dose of Study Drug | 17 | 17 | 4 | 4 | 15 | 15 | 5 | 6
Completed | 10 | 11 | 4 | 3 | 14 | 12 | 5 | 6
Not Completed | 10 | 10 | 1 | 1 | 1 | 4 | 0 | 0
Not completed — Adverse Event | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Clinical Failure | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Participant left investigator's care | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason not specified | 3 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Randomized but not treated | 3 | 4 | 1 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Vancomycin or SSP, Bacteremia, Severe Renal Impairment: Cohort 1. Participants randomized to the comparator therapy group received vancomycin or penicillinase-resistant penicillin (nafcillin, oxacillin, or cloxacillin). Investigators were allowed to select an agent based on local availability and normal treatment practices. Participants randomized to comparator subsequently found to have an infection caused by Methicillin-Susceptible Staphylococcus Aureus (MSSA) could have switched from vancomycin to penicillinase-resistant penicillin (nafcillin, oxacillin, or cloxacillin) at the Investigator's discretion. All treatments were dosed per Investigator's discretion and were administered intravenously until end of antibiotic therapy for bacteremia or until hospital discharge, whichever occurred first. Investigators treated participants according to their usual decision-making and discretion.
- Total: Total of all reporting groups
Arm/Group | Daptomycin, Bacteremia, Severe Renal Impairment | Vancomycin or SSP, Bacteremia, Severe Renal Impairment | Daptomycin, Bacteremia, Moderate Renal Impairment | Vancomycin or SSP, Bacteremia, Moderate Renal Impairment | Daptomycin, cSSSI, Severe Renal Impairment | Vancomycin or SSP, cSSSI, Severe Renal Impairment | Daptomycin, cSSSI, Moderate Renal Impairment | Vancomycin or SSP, cSSSI, Moderate Renal Impairment | Total
Number analyzed (Participants) | 17 | 17 | 4 | 4 | 15 | 15 | 5 | 6 | 83
Age, Categorical [Count of Participants; unit: Participants]
  LTE18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BTWN | 14 | 12 | 1 | 3 | 11 | 11 | 1 | 3 | 56
  GTE65 | 3 | 5 | 3 | 1 | 4 | 4 | 4 | 3 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 2 | 2 | 5 | 3 | 3 | 1 | 28
  Male | 10 | 12 | 2 | 2 | 10 | 12 | 2 | 5 | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Creatine Phosphokinase (CPK) Elevations Through End of Therapy/Early Termination (EOT/ET)
Description: The number of participants with CPK elevations of >500 units per liter (U/L) above baseline at any time from Day 1 through the EOT/ET visit are presented.
Time Frame: Baseline through EOT/ET
Population: Participants who received at least 1 dose of study drug and had a baseline CPK value and at least 1 post-baseline CPK assessment between Day 1 post-dosing and EOT visit.
Measure: Number; unit: participants
Arm/Group | Daptomycin, Bacteremia, Severe Renal Impairment | Vancomycin or SSP, Bacteremia, Severe Renal Impairment | Daptomycin, Bacteremia, Moderate Renal Impairment | Vancomycin or SSP, Bacteremia, Moderate Renal Impairment | Daptomycin, cSSSI, Severe Renal Impairment | Vancomycin or SSP, cSSSI, Severe Renal Impairment | Daptomycin, cSSSI, Moderate Renal Impairment | Vancomycin or SSP, cSSSI, Moderate Renal Impairment
Number analyzed (Participants) | 16 | 14 | 3 | 4 | 14 | 13 | 5 | 4
participants | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0

2. Secondary Outcome: Overall Therapeutic Outcome at Test of Cure (TOC)/Safety Visit
Description: Participants were assigned a Sponsor-assessed clinical outcome based on the following definitions at the TOC/Safety visit:
  Failure: Assessed as a failure at any time by the Investigator or received non-study antimicrobial therapy for lack of efficacy or had the primary site of infection removed completely by surgery or underwent surgery to treat the infection >4 days after starting study medication.
  Success: Were not assessed as a failure at any time and were assessed as a cure or improvement by the Investigator at the TOC visit.
  Non-evaluable: Received potentially effective antimicrobial therapy during the study period for reasons other than lack of efficacy or received <4 days of study medication or were not assessed by the Investigator.
Time Frame: Baseline through TOC/Safety Visit
Population: Participants who received at least 1 dose of study drug and had at least 1 Gram-positive baseline infecting pathogen for cSSSI participants or S. aureus bacteremia for bacteremia participants.
Measure: Number; unit: participants
Arm/Group | Daptomycin, Bacteremia, Severe Renal Impairment | Vancomycin or SSP, Bacteremia, Severe Renal Impairment | Daptomycin, Bacteremia, Moderate Renal Impairment | Vancomycin or SSP, Bacteremia, Moderate Renal Impairment | Daptomycin, cSSSI, Severe Renal Impairment | Vancomycin or SSP, cSSSI, Severe Renal Impairment | Daptomycin, cSSSI, Moderate Renal Impairment | Vancomycin or SSP, cSSSI, Moderate Renal Impairment
Number analyzed (Participants) | 15 | 16 | 4 | 4 | 15 | 15 | 5 | 6
participants
  Success | 9 | 9 | 1 | 3 | 10 | 9 | 5 | 4
  Failure | 2 | 1 | 2 | 0 | 3 | 2 | 0 | 2
  Non-evaluable | 4 | 6 | 1 | 1 | 2 | 4 | 0 | 0

ADVERSE EVENTS:
Groups:
- Daptomycin, Bacteremia, Severe Renal Impairment: Cohort 1. Daptomycin was given intravenously 6 milligrams per kilogram (mg/kg) per administration. For bacteremia participants with Creatinine Clearance (CLcr) below 30 milliliters per minute (mL/min) and currently receiving hemodialysis, daptomycin was administered immediately following each hemodialysis session (3 per week) for 14 to 42 days based on disease resolution or Investigator discretion. For participants not receiving dialysis, daptomycin was administered every 48 hours for 14 to 42 days based on disease resolution or Investigator discretion.)
Arm/Group | Daptomycin, Bacteremia, Severe Renal Impairment | Vancomycin or SSP, Bacteremia, Severe Renal Impairment | Daptomycin, Bacteremia, Moderate Renal Impairment | Vancomycin or SSP, Bacteremia, Moderate Renal Impairment | Daptomycin, cSSSI, Severe Renal Impairment | Vancomycin or SSP, cSSSI, Severe Renal Impairment | Daptomycin, cSSSI, Moderate Renal Impairment | Vancomycin or SSP, cSSSI, Moderate Renal Impairment
Serious Adverse Events (participants affected / at risk) | 2/17 | 6/17 | 2/4 | 1/4 | 1/15 | 5/15 | 0/5 | 2/6
Other Adverse Events (participants affected / at risk) | 9/17 | 15/17 | 4/4 | 4/4 | 4/15 | 5/15 | 2/5 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daptomycin, Bacteremia, Severe Renal Impairment (N=17) | Vancomycin or SSP, Bacteremia, Severe Renal Impairment (N=17) | Daptomycin, Bacteremia, Moderate Renal Impairment (N=4) | Vancomycin or SSP, Bacteremia, Moderate Renal Impairment (N=4) | Daptomycin, cSSSI, Severe Renal Impairment (N=15) | Vancomycin or SSP, cSSSI, Severe Renal Impairment (N=15) | Daptomycin, cSSSI, Moderate Renal Impairment (N=5) | Vancomycin or SSP, cSSSI, Moderate Renal Impairment (N=6)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Resulted in one participant death.
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Resulted in one participant death.
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Graft infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Graft complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombolysis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daptomycin, Bacteremia, Severe Renal Impairment (N=17) | Vancomycin or SSP, Bacteremia, Severe Renal Impairment (N=17) | Daptomycin, Bacteremia, Moderate Renal Impairment (N=4) | Vancomycin or SSP, Bacteremia, Moderate Renal Impairment (N=4) | Daptomycin, cSSSI, Severe Renal Impairment (N=15) | Vancomycin or SSP, cSSSI, Severe Renal Impairment (N=15) | Daptomycin, cSSSI, Moderate Renal Impairment (N=5) | Vancomycin or SSP, cSSSI, Moderate Renal Impairment (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 3 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device leakage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device complication (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenderness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis in device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest wall abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cardiac murmur (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart sounds abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (4) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin chapped (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication is initiated by Cubist. If first publication not published within 1 year of study conclusion or termination, Investigator has right to publish and disclose the data. Prior to any submission for publication, presentation, or communication of results or information arising from the study, Investigator shall provide Cubist at least 90 days for review and comment upon the manuscript or other material for such publication or presentation.